CLINICAL TRIAL: NCT03636425
Title: Prevalence of Musculoskeletal Disorders in Mountain Runners
Brief Title: Musculoskeletal Disorders in Mountain Runners
Status: Completed | Type: Observational
Sponsor: University of Bologna (Other)
Responsible Party: Principal Investigator, Paolo Pillastrini, Clinical Professor, University of Bologna
Other Study IDs: 07082018
Record Dates: First submitted 2018-08-12; First posted 2018-08-17 (Actual); Last update posted 2019-02-11 (Actual); Status verified 2019-02

CONDITIONS: Musculoskeletal Diseases
Keywords: Running; Resistance Training; Mountain; Physiotherapy
MeSH Terms: conditions — Musculoskeletal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Questionnaire administration to gather information — In the questionnaire there are questions about the training (number of kilometers traveled by runners on average, total height difference, number of training sessions per week, training ground) questions on other activities carried out (gym, bicycle, etc.) number of competitions that runners participated in the month, used footwear, musculoskeletal disorders in the last 12 months, which health professional the runner has addressed, which physiotherapy therapies did.

SUMMARY:
the study aims to estimate the prevalence of musculoskeletal disorders in a population of runners in the mountains; moreover it proposes to explore the relationship between distance traveled, the difference in height, the training frequency in the week, the shoes worn, the training method, the use of supports and experience of running with musculoskeletal disorders. The secondary objectives of this study are to investigate to which rehabilitative figures the sportsman turns and if the treatments have positive outcomes.

DETAILED DESCRIPTION:
Running is one of the most popular forms of exercise in the world. The prevalence of musculoskeletal disorders in street runners has already been extensively studied and is about 55% of those affected. In recent years, more and more runners paid their attention to mountain running where, the different types of terrain and the important differences in height require a different musculoskeletal effort. In the literature there are few studies that have investigated the prevalence of disorders, risk factors and protective factors on these runners. The mountain running performed with regularity and method is certainly a healthy activity for individuals, but it is not free from injuries due to several factors, such as long distance, significant differences in level and uneven terrain. It is not clear whether these factors can influence the onset of skeletal muscle disorders. The study aims to estimate the prevalence of musculoskeletal disorders in this population of mountain runners; moreover it proposes to explore in this population the relationship between distance traveled, the difference in height, the training frequency in the week, the shoes worn, the training method, the use of supports and experience of running with musculoskeletal disorders. Moreover, the study wants to investigate to which rehabilitative figures the sportsman turns and if the treatments have positive outcomes. Inclusion criteria are: age over 18, be a participant of at least one trail, understand the Italian language, to have signed informed consent. Recruitment: all participants in mountain races will be invited to reply to the attached questionnaire anonymously when the race bib is picked up. The runners will be free to participate or not in the survey, without the choice can affect the results of the race in any way and can create situations of subjection to the organization.

ELIGIBILITY:
Inclusion Criteria:

* age over 18,
* be a participant of at least one mountain race
* understand the Italian language
* have signed an informed consent

Exclusion Criteria:

* under the age of 18
* do not understand Italian language
* not having given consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: mountain runners participating in competitions over the age of 18
Sampling Method: Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-08-30 (Actual); Primary Completion 2019-01-20 (Actual); Study Completion 2019-01-30 (Actual)

PRIMARY OUTCOMES:
presence of musculoskeletal disorders | through study completion, an average of 6 months
  this outcome is self-reported

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Pillastrini, Principal Investigator — Bologna University
Locations (1):
- University of Bologna, Bologna, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No